CLINICAL TRIAL: NCT03697603
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled, Parallel Group-comparison Trial to Assess the Efficacy and Safety of Brexpiprazole as Adjunctive Therapy in Patients With Major Depressive Disorder
Brief Title: A Study of Brexpiprazole in Patients With Major Depressive Disorder
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 331-102-00058
Record Dates: First submitted 2018-07-24; First posted 2018-10-05 (Actual); Results first posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-03

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — brexpiprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Brexpiprazole 1mg (Experimental): Tablets, Oral, 1mg once daily, 14 weeks Other Name: REXULTI
  Interventions: Drug: Brexpiprazole
- Brexpiprazole 2mg (Experimental): Tablets, Oral, 2 mg once daily, 14 weeks Other Name: REXULTI
  Interventions: Drug: Brexpiprazole
- Placebo (Placebo Comparator): Tablets, Oral, once daily, 14 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Brexpiprazole — Tablets, Oral, once daily, 14 weeks
  Other Names: REXULTI
  Arms: Brexpiprazole 1mg; Brexpiprazole 2mg
Drug: Placebo — Tablets, Oral, once daily, 14 weeks
  Arms: Placebo

SUMMARY:
The purpose of this 14 week, randomized, double-blind, placebo controlled study is to assess the safety and efficacy of brexipiprazole to placebo as adjunctive treatment to an assigned open-label marketed antidepressant therapy (ADT) in patients with Major Depressive Disorder.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients, or inpatients at the time of informed consent whose treatment status can be successfully shifted to outpatient status before enrollment in the antidepressant treatment period
* Male and female patients ≥ 20 to < 65 years of age (at the time of informed consent)
* Patients who have a level of comprehension sufficient to allow them to give written informed consent to all of the observation/examination/evaluation items specified in the protocol, and who can understand the contents of the trial
* Patients with a DSM-5 classification-based diagnosis of "major depressive disorder, single episode" or "major depressive disorder, recurrent episode," and whose current episode has persisted for at least 8 weeks

Exclusion Criteria:

* Women who are pregnant or breastfeeding or who have positive pregnancy test (urine) results at screening
* Sexually active male subjects or sexually active female subjects of childbearing potential, who will not agree to practice 2 different methods of birth control or to remain abstinent during the trial and for 30 days after the final

IMP administration. For birth control, 2 of the following methods must be used:

vasectomy, tubal ligation, vaginal diaphragm, intra-uterine contraceptive device (IUD), oral contraceptives, or condom with spermicide.

* Patients with a treatment history showing that all antidepressants (including those not used for the current major depressive episode) cannot be tolerated
* Patients with a history of electroconvulsive therapy
* Patients with a diagnosis of any of the following diseases according to DSM-5

  1. Neurocognitive disorders
  2. Schizophrenia spectrum and other psychotic disorders
  3. Bipolar and related disorders
  4. Feeding and eating disorders
  5. Obsessive-compulsive disorder
  6. Panic disorder
  7. Posttraumatic stress disorder

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 740 (Actual)
Dates: Start 2018-07-30 (Actual); Primary Completion 2022-06-06 (Actual); Study Completion 2022-07-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nanko-kokorono clinic, Fukushima, Japan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article Publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on an Otsuka-owned remotely accessible data sharing platform with Python and R analytical software. Research requests should be directed to clinicaltransparency@Otsuka-us.com.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted in 740 participants from 145 trial sites in Japan.
Pre-assignment Details: Adults with major depressive disorder as defined by Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) and who had not responded sufficiently to antidepressants (SSRIs or SNRIs) were included.
Groups:
- Brexpiprazole 1 mg: Participants received brexpiprazole 1 mg tablet once daily for 6 weeks.
- Brexpiprazole 2 mg: Participants received brexpiprazole 1 mg tablet once daily for 1 week followed by 2 mg tablet once daily for 5 weeks.
- Placebo: Participants received placebo tablet once daily for 6 weeks.
Period: Overall Study
Arm/Group | Brexpiprazole 1 mg | Brexpiprazole 2 mg | Placebo
Started | 250 | 246 | 244
Completed | 238 | 219 | 232
Not Completed | 12 | 27 | 12
Not completed — Adverse Event | 3 | 18 | 3
Not completed — Physician Decision | 1 | 0 | 2
Not completed — Protocol Violation | 3 | 8 | 5
Not completed — Withdrawal by Subject | 5 | 1 | 1
Not completed — Protocol Violation | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) which comprised subjects who, after randomization, had received at least 1 dose of the study medication in the double-blind period (Phase B), and from whose the Montgomery Åsberg Depression Rating Scale (MADRS) total scores had been obtained at baseline and at least 1 time point after initiation of the treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Brexpiprazole 1 mg | Brexpiprazole 2 mg | Placebo | Total
Number analyzed (Participants) | 248 | 245 | 243 | 736
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 248 | 245 | 243 | 736
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.9 (10.8) | 40.0 (10.7) | 39.8 (10.8) | 40.2 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116 | 102 | 105 | 323
  Male | 132 | 143 | 138 | 413
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 248 | 245 | 243 | 736
Region of Enrollment [Number; unit: participants]
  Japan | 248 | 245 | 243 | 736

OUTCOME MEASURES:

1. Primary Outcome: Mean Changes From Baseline (Week 8 of the Antidepressant Treatment Period [Phase A]) in the MADRS Total Scores at Week 6 of the Double-blind Period (Phase B).
Description: The MADRS was a clinician-rated scale which evaluated the level of depression. The MADRS consisted of 10 items assessing apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, suicidal thought. Each item was scored from 0 to 6, with higher scores indicating worse condition. Summed subscales were combined to compute a total score. Total score ranges from 0 to 60, with higher scores indicating worse condition.The mean changes were compared between antidepressant treatments and brexpiprazole as adjunctive therapy.
Time Frame: Baseline (the end of Phase A), at completion of administration (Week 6).
Population: FAS (Same as Baseline Analysis Population Description)
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole 1 mg | Brexpiprazole 2 mg | Placebo
Number analyzed (Participants) | 248 | 245 | 243
Units on a scale | -8.5 (0.47) | -8.2 (0.47) | -6.7 (0.47)
Statistical Analysis 1: Comparison: Brexpiprazole 2 mg vs Placebo; Statistical analysis to compare brexpiprazole 2 mg/day and placebo was performed at Week 6; Test type: Superiority; p = 0.0312, MMRM; Mean Difference (Final Values) = -1.4, 95% CI 2-sided [-2.7 to -0.1]
Statistical Analysis 2: Comparison: Brexpiprazole 1 mg vs Placebo; Statistical analysis to compare brexpiprazole 1 mg/day and placebo was performed at Week 6; Test type: Superiority; p = 0.0089, MMRM; Mean Difference (Final Values) = -1.7, 95% CI 2-sided [-3.0 to -0.4]

2. Secondary Outcome: CGI-I Improvement Rate at Week 6 of the Double-blind Period (Phase B)
Description: Clinical Global Impression - Improvement (CGI-I) improvement rate: the proportion of participants who score 1 or 2 on the CGI-I scale at Week 6 of the double-blind period (Phase B).
  The CGI-I Scale was a clinician-rated scale which assessed the total improvement of the participant's condition compared to that at baseline. Scores range from 0 to 7:0 = Not assessed, 1= Very much improved, 2 = Much improved, 3= Minimally improved, 4= No change, 5= Minimally worse, 6= Much worse, 7= Very much worse. Higher scores indicated worse condition.
Time Frame: Baseline (the end of Phase A), at completion of administration (Week 6).
Population: FAS (Same as Baseline Analysis Population Description)
Measure: Number; unit: percentage of participants
Arm/Group | Brexpiprazole 1 mg | Brexpiprazole 2 mg | Placebo
Number analyzed (Participants) | 248 | 245 | 243
percentage of participants | 35.1 | 35.1 | 29.6
Statistical Analysis 1: Comparison: Brexpiprazole 2 mg vs Placebo; Statistical analysis to compare brexpiprazole 2 mg/day and placebo was performed at Week 6; Test type: Other; p = 0.1964, Chi-squared; Diff = 5.5, 95% CI 2-sided [-2.8 to 13.8]
Statistical Analysis 2: Comparison: Brexpiprazole 1 mg vs Placebo; Statistical analysis to compare brexpiprazole 1 mg/day and placebo was performed at Week 6; Test type: Other; p = 0.1969, Chi-squared; Diff = 5.5, 95% CI 2-sided [-2.8 to 13.7]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from signing of the informed consent form until post-treatment observation period for up to 30 days (±5 days) after the final day of study medication administration (end of trial date [final day of observation]).
Description: Subjects who received at least one dose of IMP were included in the safety analysis.
Arm/Group | Brexpiprazole 1 mg | Brexpiprazole 2 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/250 | 0/246 | 0/244
Serious Adverse Events (participants affected / at risk) | 3/250 | 3/246 | 2/244
Other Adverse Events (participants affected / at risk) | 108/250 | 153/246 | 92/244
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brexpiprazole 1 mg (N=250) | Brexpiprazole 2 mg (N=246) | Placebo (N=244)
Alcoholic pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Extramammary Paget's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 1 | 0
IIIrd nerve paralysis (Nervous system disorders) | 1 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brexpiprazole 1 mg (N=250) | Brexpiprazole 2 mg (N=246) | Placebo (N=244)
Hyperprolactinaemia (Endocrine disorders) | 3 | 13 | 3
Constipation (Gastrointestinal disorders) | 5 | 9 | 5
Diarrhoea (Gastrointestinal disorders) | 6 | 7 | 7
Nausea (Gastrointestinal disorders) | 1 | 8 | 6
Salivary hypersecretion (Gastrointestinal disorders) | 2 | 6 | 1
Malaise (General disorders) | 1 | 7 | 2
Pyrexia (General disorders) | 7 | 1 | 6
Hepatic function abnormal (Hepatobiliary disorders) | 3 | 8 | 6
Nasopharyngitis (Infections and infestations) | 20 | 16 | 24
Alanine aminotransferase increased (Investigations) | 8 | 7 | 4
Aspartate aminotransferase increased (Investigations) | 6 | 4 | 3
Blood creatine phosphokinase increased (Investigations) | 2 | 9 | 5
Blood insulin increased (Investigations) | 5 | 6 | 1
Blood prolactin increased (Investigations) | 6 | 15 | 6
Gamma-glutamyltransferase increased (Investigations) | 6 | 3 | 3
Weight increased (Investigations) | 18 | 19 | 6
Increased appetite (Metabolism and nutrition disorders) | 3 | 6 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 5 | 4
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 3 | 5 | 1
Akathisia (Nervous system disorders) | 15 | 60 | 3
Dizziness (Nervous system disorders) | 4 | 5 | 6
Extrapyramidal disorder (Nervous system disorders) | 1 | 11 | 2
Headache (Nervous system disorders) | 6 | 3 | 11
Somnolence (Nervous system disorders) | 3 | 8 | 6
Tremor (Nervous system disorders) | 16 | 12 | 9
Insomnia (Psychiatric disorders) | 9 | 12 | 8
Hypertension (Vascular disorders) | 8 | 6 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-01-23): https://cdn.clinicaltrials.gov/large-docs/03/NCT03697603/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-10): https://cdn.clinicaltrials.gov/large-docs/03/NCT03697603/SAP_001.pdf